CLINICAL TRIAL: NCT04005066
Title: A Post-Marketing Clinical Study to Evaluate the Safety of Elunate® (Fruquintinib Capsules) in Chinese Patients.
Brief Title: A Phase IV Study of Elunate® (Fruquintinib) in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-013-00CH2
Record Dates: First submitted 2019-04-18; First posted 2019-07-02 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Patient Safety
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: * Currently using Elunate® or will use Elunate®(Fruquintinib) within a week;
  * Provision of informed consent by the patient.
  Interventions: Drug: Elunate®

INTERVENTIONS:
Drug: Elunate® — The recommended dose is 5 mg once daily (1 capsule, each capsule contains 5 mg of fruquintinib); three weeks of continuous drug administration followed by one week of drug free period (4 weeks as one treatment cycle).
  Other Names: Fruquintinib

SUMMARY:
A phase IV study to characterize safety of Elunate® (Fruquintinib) in Chinese patients

DETAILED DESCRIPTION:
This study is a prospective, open-label, multi-center, study design to obtain the safety information of participant after medication. The follow-up time points for each participant include first time signing the informed consent form,1 month after signing the informed consent form, 6 months after signing the informed consent form or 30 days after the last dose (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Currently using Elunate®(Fruquintinib) or will use Elunate®(Fruquintinib) within a week;
* Provision of informed consent by the patient.

Exclusion Criteria:

• Unsuitable for the study according to investigator's judgement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Advanced solid tumor patients treated with Elunate®( fruquintinib) in Chinese real world practice
Sampling Method: Non-Probability Sample
Enrollment: 3005 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs | from the first administration of fruquintinib up to 6 months
  % of patients with AEs according to CTCAE 4.03
Incidence of ADRs | from the first administration of fruquintinib up to 6 months
  % of patients with ADRs according to CTCAE 4.03
Incidence of SAEs | from the first administration of fruquintinib up to 6 months
  % of patients with SAEs according to CTC AE 4.03
Incidence of AESI | from the first administration of fruquintinib up to 6 months
  % of patients with AESI according to CTC AE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Xue, Study Director — Hutchmed
Locations (1):
- Shanghai Dongfang Hospital, Shanghai, China